CLINICAL TRIAL: NCT03408990
Title: Confounding Factors of Impedance Pneumography Signal Changes During Sleep
Brief Title: Confounding Factors of Impedance Pneumography
Status: Completed | Type: Observational
Sponsor: Revenio Research (Industry)
Collaborators: Children's Hospital Srebrnjak (Other)
Responsible Party: Sponsor
Other Study IDs: VCS-005
Record Dates: First submitted 2018-01-16; First posted 2018-01-24 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Healthy; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep study for clinical reasons: Children referred to sleep study for clinical reasons
- Healthy: Healthy children, no relevant pathologies

SUMMARY:
The purpose of this study is to evaluate the association of signals recorded and analysed with Ventica® Lung Function Testing System (LFTS) in infants and pre-schoolers during the whole night sleep with the gold standard for sleep recording events, polysomnography, in order to better understand the confounding factors for momentary changes in the impedance pneumography-derived tidal breathing flow-volume (TBFV) curves.

ELIGIBILITY:
Group 1: (children referred to sleep study for clinical reasons) Inclusion criteria:

* Age 1-7 years, both sexes
* Referred to polysomnography
* Signed informed consent

Group 2: (healthy children) Inclusion criteria:

* 2-7 years, both sexes
* Healthy at the time of inclusion based on history and clinical examination according to the investigator judgement
* Lung function in the reference range
* Signed informed consent

Exclusion Criteria:

* Preterm birth with chronic respiratory disorder of prematurity
* Significant nasal congestion or adenotonsillar hypertrophy with signs and symptoms of sleep apnea or sleep disordered breathing
* Chronic rhinosinusitis, synonasal polyposis
* Personal or family history or clinical evidence of asthma, atopy or other chronic respiratory disorders (high risk for asthma and allergy)
* Use of asthma rescue or maintenance medication within 4 weeks prior to inclusion
* Recurrent bronchitis or recurrent hospitalizations because of a respiratory illness (recurrent pneumonia)
* Hospital-treated for bronchiolitis with residual symptoms
* Acute respiratory infection or hospitalization because of an acute illness within 4 weeks prior to inclusion
* Other cardiorespiratory or neurological chronic diseases or states that may significantly alter the overnight breathing pattern
* Implanted or external active medical devices
* Long lasting respiratory events during the polysomnography study like continuous upper airway limitation

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Subjects referred to sleep laboratory at the investigational site or healthy volunteers from Zagreb and surroundings
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Association between sleep stages and tidal breathing flow-volume (TBFV) curves | 1 night
  Assess the correlation between Ventica-derived TBFV curves within and between different EEG-derived sleep stages during night sleep

SECONDARY OUTCOMES:
Association between body/head positions and tidal breathing flow-volume (TBFV) curves | 1 night
  Assess the correlation between Ventica-derived TBFV curves within and between different body/head positions (derived from video and/or positional sensors) during night sleep

CONTACTS AND LOCATIONS:
Overall Officials: Davor Plavec, MD, PhD, Principal Investigator — Children's Hospital Srebrnjak
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No